CLINICAL TRIAL: NCT03693404
Title: Effects of a Surgical Site Injection on Pain Scores and Narcotic Use After Orthopaedic Trauma Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-01019
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Results first posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-06

CONDITIONS: Pertrochanteric Fracture
MeSH Terms: interventions — Bupivacaine; Morphine; Ketorolac; Anesthetics, General

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spinal Anesthesia (Experimental): Injection of 40cc 0.25% Marcaine, 5 mg Duramorph (1 mg/cc, 5 cc total), and 30 mg of ketorolac (30 mg/cc, 1 cc total) into the periosteum, and musculature surrounding the fracture site and 0.25% Bupivacaine (Marcaine) 10 mL into the subcutaneous tissue surrounding the surgical incision.
  Interventions: Drug: Marcaine, Duramorph , ketorolac; Drug: Bupivacaine (Marcaine)
- General Anesthesia (Active Comparator): The control group will receive no injection into area surrounding the fracture site
  Interventions: Drug: General Anesthetics

INTERVENTIONS:
Drug: Marcaine, Duramorph , ketorolac — Subjects in the SSI group will receive an injection of 40cc 0.25% Marcaine, 5 mg Duramorph (1 mg/cc, 5 cc total), and 30 mg of ketorolac (30 mg/cc, 1 cc total) into the periosteum, and musculature surrounding the fracture site and 0.25% Bupivacaine (Marcaine) 10 mL into the subcutaneous tissue surrounding the surgical incision.
  Arms: Spinal Anesthesia
Drug: Bupivacaine (Marcaine) — 0.25% Bupivacaine (Marcaine) 10 mL into the subcutaneous tissue surrounding the surgical incision.
  Arms: Spinal Anesthesia
Drug: General Anesthetics — Placebo group will only receive standard of care general anesthesia
  Arms: General Anesthesia

SUMMARY:
This is a phase I, randomized, single-blind, placebo-controlled, single-center study of the effects of surgical site injection on pain and narcotic utilization in participants who undergo surgery for lower extremity fractures. 200 participants with lower extremity fractures who are admitted for operative fixation will be included in the study. Participants will be randomized to receive either a pain cocktail injection around the fracture site and surrounding tissues or control (no injection). An analysis of pain scores, rehabilitation progress, length of stay, narcotic utilization, and satisfaction scores will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Lower extremity fracture including femoral neck, intertrochanteric, sub-trochanteric, and femoral shaft fracture

Exclusion Criteria:

* Pregnant women
* Treatment with Arthroplasty
* Patients who receive a peripheral nerve block
* Patients who receive intra-op or post-op ketamine
* Patients with concomitant TBI or MR
* Polytrauma patients
* Pathologic Fractures
* Patients who live greater than 10 miles from NYU or who will not be followed by an NYU provider
* Patients with a contraindication to any of the medications on the study list due to other medical problems such as renal or liver disease or due to allergy/intolerance
* Patients with prior extremity weakness resulting from stroke or other neurological condition
* Prior or current history of narcotic use
* Patients with advanced dementia
* NYUMC Students, Residents, Faculty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-06-05 (Actual); Study Completion 2021-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Leucht, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: SAP, CSR
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Requests should be directed to Philipp.Leucht@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Ihejirika-Lomedico R, Solasz S, Lorentz N, Egol KA, Leucht P; and NYU Hip Fracture Research Group. Effects of Intraoperative Local Pain Cocktail Injections on Early Function and Patient-Reported Outcomes: A Randomized Controlled Trial. J Orthop Trauma. 2023 Sep 1;37(9):433-439. doi: 10.1097/BOT.0000000000002628. PMID 37199438

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | General Anesthesia | Spinal Anesthesia
Started | 109 | 81
Completed | 108 | 75
Not Completed | 1 | 6
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 5
Not completed — Excluded from Analysis | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | General Anesthesia | Spinal Anesthesia | Total
Number analyzed (Participants) | 109 | 75 | 184
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.5 (15.3) | 77.5 (11.6) | 76.5 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 47 | 123
  Male | 33 | 28 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 95 | 62 | 157
  More than one race | 11 | 7 | 18
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 109 | 75 | 184

OUTCOME MEASURES:

1. Primary Outcome: Amount (mg) of Narcotics (Oral Morphine mg Equivalents) Used
Description: Number of mgs taken of oral morphine
Time Frame: Post-Operative Day 0
Measure: Mean (Standard Deviation); unit: morphine milligram equivalents (MME)
Arm/Group | General Anesthesia | Spinal Anesthesia
Number analyzed (Participants) | 109 | 75
morphine milligram equivalents (MME) | 16 (1.5) | 10 (1.4)

2. Primary Outcome: Ambulation Distance
Description: Ambulation is the ability to walk without the need for any kind of assistance. It is most often used when describing the goals of a patient after a surgery or physical therapy.
Time Frame: Post-operative Day 3
Measure: Mean (Standard Deviation); unit: Feet
Arm/Group | General Anesthesia | Spinal Anesthesia
Number analyzed (Participants) | 109 | 75
Feet | 48.7 (8) | 88.9 (17.6)

3. Primary Outcome: Score on Visual Analogue Scale (VAS) for Pain
Description: VAS is a tool widely used to measure pain. A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 100 mm horizontal line, and this rating is then measured from the left edge (=VAS score). The total score range is 0 (no pain) to 10 (worst pain imaginable); the higher the score, the worse the pain.
Time Frame: Hour 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | General Anesthesia | Spinal Anesthesia
Number analyzed (Participants) | 109 | 75
score on a scale | 3.3 (1.7) | 2.5 (1.4)

ADVERSE EVENTS:
Time Frame: 3 months
Description: regular investigator assessment / questionnaire
Arm/Group | General Anesthesia | Spinal Anesthesia
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/81
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/81
Other Adverse Events (participants affected / at risk) | 0/109 | 0/81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/04/NCT03693404/Prot_SAP_000.pdf